CLINICAL TRIAL: NCT07345702
Title: Endovascular Versus Medical Therapy for Acute Large-Core Basilar Artery Occlusion: A Multicenter Retrospective Registry Study (BAOCHE-LC)
Brief Title: Basilar Artery Occlusion Chinese Endovascular Registry in Patients With Large-Core Infarct
Acronym: BAOCHE-LC
Status: Not yet recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Chuanhui Li, Associate Professor, Xuanwu Hospital, Captimal Medical University, Xuanwu Hospital, Beijing
Other Study IDs: BAOCHE-LC
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Basilar Artery Occlusion; Ischemic Stroke; Large Core Infarct
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Endovascular Therapy
  Interventions: Procedure: Endovascular Therapy
- Best Medical Treatment Alone

INTERVENTIONS:
Procedure: Endovascular Therapy — Endovascular therapy performed as part of routine clinical care for acute basilar artery occlusion, including mechanical thrombectomy with stent retriever and/or aspiration. Rescue angioplasty and/or intracranial stenting may be used at the operator's discretion. Peri-procedural management and concomitant medical therapy follow local standard practice.
  Groups: Endovascular Therapy

SUMMARY:
This multicenter retrospective registry study evaluates the safety and effectiveness of endovascular therapy versus medical therapy for acute large-core basilar artery occlusion. It also investigates clinical, imaging, and laboratory factors associated with functional outcomes and mortality. Patients are grouped according to the treatment received in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, men or women.
2. Occlusion (TIMI 0-1) of the basilar artery or intracranial segments of both vertebral arteries (V4) as evidenced by CTA/MRA/DSA.
3. Time from symptom onset (or last known well) to treatment (endovascular therapy or medical therapy) ≤7 days.
4. Patients with large core infarction in the posterior circulation, defined as a posterior circulation Acute Stroke Prognosis Early CT score (pc-ASPECTS) score of 0-5 on CT angiography source images or MR with diffusion-weighted imaging or non-contrast CT.

Exclusion Criteria:

1. Subjects with occlusions in both anterior and posterior circulation.
2. CT or MR evidence of hemorrhage (the presence of microbleeds on MRI is allowed).
3. Missing key clinical information (e.g., unavailable baseline NIHSS, unclear symptom onset/last known well time, or missing major treatment information including whether EVT was performed).
4. Baseline NIHSS score <6.
5. Woman of childbearing potential who is known to be pregnant or lactating or who has a positive pregnancy test on admission.
6. Missing follow-up outcomes at 90 days.
7. Any other condition judged by investigators to substantially affect analysis or interpretation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) with imaging-confirmed acute vertebrobasilar occlusion and large-core infarction (pc-ASPECTS 0-5) treated within 7 days of symptom onset/last known well at participating centers in China. Patients are identified retrospectively from routine clinical practice and classified according to treatment received: endovascular therapy plus standard medical management versus standard medical management alone.
Sampling Method: Non-Probability Sample
Enrollment: 518 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Achieving mRS 0-3 at 90 Days | 90 days
  The modified Rankin scale (range, 0 [no symptoms] to 6 [death]). Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Ordinal Shift analysis of mRS at 90 days | 90 days
  The modified Rankin scale (range, 0 [no symptoms] to 6 [death])
Rate of All-Cause Mortality at 90 Days | 90 days
  Death from any cause within 90 days.
Rate of Symptomatic Intracranial Hemorrhage | 24 (-2/+12) hours
Proportion of Patients Achieving mRS 0-3 at 1 year | 1 year
  The modified Rankin scale (range, 0 [no symptoms] to 6 [death]). Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The study is proceeding.